CLINICAL TRIAL: NCT05558267
Title: A Randomized, Pilot, Double-Blind Crossover Trial of a Potassium Containing Salt-Substitute in Hemodialysis-Dependent End Stage Kidney Disease
Brief Title: Potassium Containing Salt-Substitute in Hemodialysis-Dependent End Stage Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 22-00769
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: End Stage Kidney Disease
Keywords: Potassium-Containing Salt Substitute
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Table Salt, then Salt Substitute (Experimental): The two intervention periods will last 16 days with a 19-day washout period in between.
  During the first 16-day treatment period, participants will receive the Standard Table Salt to use for cooking and as an additive at the table. Participants will then undergo a 19-day washout period. The second 16-day treatment period will immediately follow the washout period. During the second 16-day treatment period, participants will receive the Salt Substitute to use for cooking and as an additive at the table.
  Participants will be encouraged to replace their use of regular salt with the Standard Table Salt and Salt Substitute. They will be encouraged to reduce their overall intake of salt throughout the study period. There are no restrictions or further instructions regarding timing or dosing.
  In addition, participants will undergo standard of care hemodialysis (typically 3x/week) and have their blood chemistries measured according to the usual standard of care during the study.
  Interventions: Dietary Supplement: Standard Table Salt; Dietary Supplement: Salt Substitute
- Salt Substitute, then Standard Table Salt (Experimental): The two intervention periods will last 16 days with a 19-day washout period in between.
  During the first 16-day treatment period, participants will receive the Salt Substitute to use for cooking and as an additive at the table. Participants will then undergo a 19-day washout period. The second 16-day treatment period will immediately follow the washout period. During the second 16-day treatment period, participants will receive the Standard Table Salt to use for cooking and as an additive at the table.
  Participants will be encouraged to replace their use of regular salt with the Standard Table Salt and Salt Substitute. They will be encouraged to reduce their overall intake of salt throughout the study period. There are no restrictions or further instructions regarding timing or dosing.
  In addition, participants will undergo standard of care hemodialysis (typically 3x/week) and have their blood chemistries measured according to the usual standard of care during the study.
  Interventions: Dietary Supplement: Standard Table Salt; Dietary Supplement: Salt Substitute

INTERVENTIONS:
Dietary Supplement: Standard Table Salt — Standard Table Salt is administered orally. It is transferred to unmarked saltshakers by non-blinded research coordinators. The unmarked saltshaker is delivered to the participant during dialysis.
  Other Names: Morton Standard Table Salt
Dietary Supplement: Salt Substitute — Salt Substitute is available as a crystalized powder. It substitutes potassium chloride for sodium chloride, and thus contains about 50% less sodium than standard table salt.
  Salt Substitute is administered orally. It is transferred to unmarked saltshakers by non-blinded research coordinators. The unmarked saltshaker is delivered to the participant during dialysis.
  Other Names: Morton Lite Salt

SUMMARY:
16 individuals with hemodialysis-dependent end stage kidney disease will receive 16 days of a potassium-containing salt-substitute and 16 days of standard table salt in random order. There will be a 19 day wash out period between the salt-substitute and table salt periods. Potassium concentration will be measured bi-weekly prior to HD each week during intervention. The primary endpoint will be the change in potassium from baseline. Additional measurements will include assessment of dietary intake, ambulatory blood pressure, occurrence of peri-dialytic symptoms, and per-dialytic vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving outpatient maintenance HD therapy.
2. Age ≥ 21 years.
3. Negative serum pregnancy test for women of child-bearing capacity. Childbearing capacity will be defined by report of menstruation within ≤ 6 months.

Exclusion Criteria:

1. Currently incarcerated.
2. Insufficient capacity for informed consent.
3. Non-hemolyzed serum potassium concentration >6.0 mEq/L within ≤30 days.
4. Unscheduled HD for hyperkalemia within ≤30 days.
5. Attendance at ≤10 of last 13 scheduled OP HD sessions.
6. Co-habiting family member with known hyperkalemia.
7. Co-habiting family with ≥stage 3b chronic kidney disease or chronic kidney disease of unknown severity.
8. Hemoglobin < 8.0 mg/dL.
9. Use of other potassium supplements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Potassium Concentration During First Treatment Period | Day 1, Day 16
  Serum potassium concentration expressed in milliequivalents per liter (mEq/L).
Change in Serum Potassium Concentration During Second Treatment Period | Day 36, Day 52
  Serum potassium concentration expressed in mEq/L.

SECONDARY OUTCOMES:
Number of Participants Presenting with Severe Hyperkalemia During First Treatment Period | Up to Day 16
  Severe hyperkalemia defined as pre-dialysis potassium levels greater than 6.5 mEq/L. The first treatment period spans from Day 1 to Day 16.
Number of Participants Presenting with Severe Hyperkalemia During Second Treatment Period | From Day 36 up to Day 52
  Severe hyperkalemia defined as pre-dialysis potassium levels greater than 6.5 mEq/L. The second treatment period spans from Day 36 to Day 52.
Number of Participants Presenting with Moderate Hyperkalemia | Up to Day 52
  Moderate hyperkalemia defined as pre-dialysis potassium levels greater than 6.0 mEq/L and less than 6.5 mEq/L.
Mean Potassium Concentration During First Treatment Period | Up to Day 16
  Potassium concentration expressed in mEq/L. The first treatment period spans from Day 1 to Day 16.
Mean Potassium Concentration During Second Treatment Period | From Day 36 up to Day 52
  Potassium concentration expressed in mEq/L. The second treatment period spans from Day 36 to Day 52.
Change in Ambulatory Systolic Blood Pressure During First Treatment Period | Day 1, Day 16
  Ambulatory systolic blood pressure expressed in millimeters of mercury (mm Hg).
Change in Ambulatory Systolic Blood Pressure During Second Treatment Period | Day 36, Day 52
  Ambulatory systolic blood pressure expressed in mm Hg.
Mean Pre-Dialysis Systolic Blood Pressure During First Treatment Period | Up to Day 16
  Pre-dialysis systolic blood pressure expressed in mm Hg. The first treatment period spans from Day 1 to Day 16.
Mean Pre-Dialysis Systolic Blood Pressure During Second Treatment Period | From Day 36 up to Day 52.
  Pre-dialysis systolic blood pressure expressed in mm Hg. The second treatment period spans from Day 36 to Day 52.
Number of Participants Presenting with Intradialytic Hypotension | Up to Day 52
  Intradialytic hypotension defined as a systolic blood pressure of less than 100 mmHg or a systolic blood pressure decrease of greater than 10 mmHg, or a mean arterial pressure decrease of greater than 30 mmHg with or without symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD MSc, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David Charytan, MD MSc (David.charytan@Nyulangone.org). The protocol will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to David.charytan@Nyulangone.org. To gain access, data requestors will need to sign a data access agreement.